CLINICAL TRIAL: NCT01056679
Title: Phase I Trial of AVD Plus Lenalidomide (Revlimid) in Elderly Intermediate or Advanced Stage Hodgkin Lymphoma Patients
Brief Title: Adriamycin, Vinblastine, DTIC and Revlimid in Elderly Hodgkin Lymphoma Patients
Acronym: AVD-Rev
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Cologne (Other)
Responsible Party: Principal Investigator, Prof. Dr. Andreas Engert, Prof., University of Cologne
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AVD-Rev
Record Dates: First submitted 2009-09-08; First posted 2010-01-26 (Estimated); Last update posted 2018-03-22 (Actual); Status verified 2018-03

CONDITIONS: Hodgkin Lymphoma
MeSH Terms: conditions — Hodgkin Disease | interventions — Doxorubicin; Dacarbazine; Lenalidomide; Vinblastine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- AVD-Rev (Experimental): Patients with intermediate stage HL receive 4 cycles of AVD-Rev followed by 30 Gy IF-RT Patientes with advanced stage HL receive 6 to 8 cycles of AVD-Rev followed by 30 GY IF-RT depending on the FDG-PET results
  Interventions: Drug: Doxorubicine; Drug: DTIC; Drug: Lenalidomide; Drug: Vinblastine

INTERVENTIONS:
Drug: Doxorubicine — 50mg/m2 day 1 + 15
Drug: DTIC — 375mg/m2 day 1 + 15
Drug: Lenalidomide — day 1 - 21
Drug: Vinblastine — 6mg/m2 day 1 + 15

SUMMARY:
The purpose of this study is to determine within the scope of the trial what the maximum tolerated dose (MTD) of lenalidomide in combination with AVD should be.

ELIGIBILITY:
Inclusion Criteria:

* Hodgkin Lymphoma, intermediate or advanced stage
* Age >60 and <75 years
* ECOG 2 or better
* No major organ dysfunction
* Ability to take aspirin or LMW Heparin

Exclusion Criteria:

* HL as composite lymphoma
* Prior use of lenalidomide
* Prior use of chemo- or radiotherapy

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2010-04; Primary Completion 2014-04 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Dose limiting toxicities (DLT)

SECONDARY OUTCOMES:
Overall response rate (ORR)
Progression free survival (PFS) | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Engert, Prof., Principal Investigator — University of Cologne
Locations (1):
- 1st Dept. of Medicine, Cologne University Hospital, Cologne, North Rhine-Westphalia, Germany

REFERENCES:
- See also: Related Info — http://www.ghsg.org